CLINICAL TRIAL: NCT05700149
Title: Integrated Molecular and Clinical Profiling to Improve Disease Characterization and Outcome Prediction in Nodal Marginal Zone Lymphoma
Status: Recruiting | Type: Observational
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Other Study IDs: IELSG52
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Nodal Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor biological material of patients with diagnosis of NMZL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
International retrospective observational cohort study aimed to describe a molecular classification for NMZL.

DETAILED DESCRIPTION:
Already existing and coded tumor biological material and health-related patient data will be retrospectively collected from institutional biobanks and patients' charts or electronic medical records upon receipt of ethical approval. Each patient enrolled in the study will be assigned to a unique identification numerical code upon registration in the study. The unique identification code will be used to record health-related data and to label biological samples. The coded biological material will be transferred to the coordinating center at the Oncology Institute of Southern Switzerland and Institute of Oncology Research in Bellinzona. Health-related data will be collected in the eCRF (OpenClinica). Data quality will be insured by query generation.

Annotated baseline features will include date of diagnosis, date of lymph node biopsy, age, gender, ECOG PS, Ann Arbor stage, LDH, number and location of extranodal sites, bone marrow involvement and percentage, peripheral blood involvement, number of nodal sites, B symptoms, lymph nodes larger than 7 cm, Hb, platelets, lymphocytes, beta-2-microglobulin, albumin, HCV infection, serum paraprotein and type.

Annotated follow-up features included date of progression to a disease requiring treatment, type of first line treatment, date of start of first line treatment, date of progression after first line treatment, date of second line treatment, type of second line treatment, date of transformation, date of death, cause of death, date of last follow-up.

Mutation analysis, immunoglobulin gene rearrangement analysis, copy number aberration analysis, structural variant analysis and DNA methylation profile will be performed by next generation sequencing of genomic DNA extracted from the lymph node biopsy. Gene expression will be assessed by next generation sequencing of RNA extracted from the lymph node biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults 18 years or older
2. Diagnosis of NMZL on lymph node histology after Jan 1st, 2000
3. Availability of tumor material from lymph node (either frozen or FFPE) collected when the patient was treatment naïve
4. Availability of the baseline and follow-up annotations

Exclusion Criteria:

1. Nodal spread of a clinically occult extranodal MZL (this must have been ruled out by carefully evaluating the extranodal tissues draining to the involved lymph nodes by imaging or endoscopy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of NMZL on lymph node histology
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Define and quantify molecular subsets. | Two years: from the end of samples collection to the end of study analysis

CONTACTS AND LOCATIONS:
Overall Officials: Davide Rossi, MD, Study Chair — Oncology Institute of Southern Switzerland and Institute of Oncology Research
Locations (36):
- United States (2):
  - University of Miami, Miami, Florida
  - Weill Cornell Medical, New York, New York
- Hematology Center after Prof. Yeolyan, Yerevan, Armenia
- University Hospital Centre Zagreb, Zagreb, Croatia
- Italy (22):
  - AO SS Antonio e Biagio e C. Arrigo, Alessandria, AL
  - Istituto Tumori "Giovanni Paolo II" I.R.C.C.S., Bari, BA
  - ASST Papa Giovanni XXIII, Bergamo, BG
  - ASST degli Spedali Civili di Brescia, Brescia, BS
  - AOU Policlinico Vittorio Emanuele, Presidio Ferrarotto, Catania, CT
  - Azienda Ospedaliero Universitaria di Ferrara, Cona, FE
  - Azienda Ospedaliera Universitaria Careggi, Florence, FI
  - Azienda Ospedaliera Papardo, Messina, ME
  - IRCCS Ospedale San Raffaele, Milan, MI
  - IEO Istituto Europeo di Oncologia, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Azienda Sanitaria Locale di Pescara, Pescara, PE
  - Centro di Riferimento Oncologico, Aviano, PN
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - AUSL IRCCS di Reggio Emilia, Arcispedale S. Maria Nuova, Reggio Emilia, RE
  - Fondazione PTV - Policlinico Tor Vergata, Rome, RM
  - Sapienza University - AOU Policlinico Umberto I, Rome, RM
  - Fondazione Policlinico Univeristario A. Gemelli, IRCCS, Università Cattolica S. Cuore, Rome, RM
  - ASST dei Sette Laghi - Ospedale di Circolo di Varese, Varese, VA
  - IRCCS - Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - AOU Maggiore della Carità, Novara
- Portuguese Institute of Oncology, Lisbon, Portugal
- Chonnam National University Hwasun Hospital, Hwasun-gun, South Korea
- Switzerland (5):
  - University Hospital Basel, Basel
  - Oncology Institute of Southern Switzerland and Institute of Oncology Research, Bellinzona
  - Hôpitaux Universitaires Genevois, Geneva
  - Kantonsspital St. Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich
- United Kingdom (3):
  - Leicester Royal Infirmary, Leicester
  - Norfolk and Norwich University Hospital, Norwich
  - Oxford University Hospitals, Oxford